CLINICAL TRIAL: NCT03169426
Title: Effect of Beta-blocker on Cardioprotective Effect of Remote Ischemic Conditioning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB_RIPC
Record Dates: First submitted 2017-05-16; First posted 2017-05-30 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Myocardial Infarction
Keywords: remote ischemic conditioning; beta-blocker
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta Blockers Carvedilol Phosphate (Experimental): Subjects are going to take beta-blocker (carvedilol, 12.5 mg once) before undergoing remote ischemic conditioning.
  Intervention: taking beta-blocker
  Interventions: Drug: Beta Blockers Carvedilol Phosphate
- Control (No Intervention): Subjects are going to undergo remote ischemic conditioning without taking any drug.

INTERVENTIONS:
Drug: Beta Blockers Carvedilol Phosphate — Subjects are going to take Beta Blockers Carvedilol Phosphate (12.5mg once) before undergoing remote ischemic conditioning.
  Arms: Beta Blockers Carvedilol Phosphate

SUMMARY:
Remote ischemic conditioning has been shown to protect myocardium from ischemia-reperfusion injury during cardiac intervention or cardiac surgery. However, effect of beta-blocker, commonly used cardiovascular medication in patients with cardiac diseases such as hypertension or angina pectoris, on cardioprotective role of remote ischemic conditioning has not been well documented. The purpose of the study is to investigate the effect of beta-blocker on remote ischemic conditioning in healthy volunteers.

DETAILED DESCRIPTION:
This study is prospective cross-over study investigating effect of beta-blocker on cardioprotective role of remote ischemic conditioning. Eleven male healthy volunteers are going to take oral beta-blocker (carvedilol, 12.5 mg once) or not before undergoing remote ischemic conditioning (consisting of 4 cycles of 5-min ischemia and subsequent 5-min reperfusion of upper arm), separated by 6-day wash-out period. To evaluate cardioprotective effect of remote ischemic conditioning, blood samples will be obtained before and after remote ischemic conditioning. Form the samples, human dialysate will be obtained and be perfused to rat heart through Langendorff apparatus before ischemia-reperfusion injury to the rat heart. Changes of infarct size of the rat heart will be compared between the beta-blocker and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer
* Not taking any medication

Exclusion Criteria:

* BMI < 18 kg/m2 or > 30 kg/m2
* Allergic history of any medication
* Baseline SBP > 150 mmHg or < 100 mmHg
* Baseline DBP > 100 mmHg or < 50 mmHg
* Strenuous exercise, excessive caffeine or alcohol, smoking 24 h prior to experiment
* Cannot undergoing remote ischemic conditioning for any reason
* Refuse to enroll

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Changes in infarct size of rat heart perfused with human dialysate after taking beta-blocker or not to evaluate the effect of beta blocker on remote ischemic conditioning performed to healthy volunteers | 24 hour after remote ischemic conditioning to healthy volunteers
  Infarct size measurement after perfusing the rat heart with human serum-derived dialysate and comparison before and after remote ischemic conditioning performed to healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No